CLINICAL TRIAL: NCT03988478
Title: Effectiveness of Inpatient Alcohol Detoxification and Psychotherapeutic Support Program
Brief Title: Inpatient Alcohol Detox & Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Jugu Maya Chaudhary, Psychologist, Tribhuvan University, Nepal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOPMH-Inpt-detox-Psychotherapy
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Inactivation, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral, detoxificaiton & psychotherapy (Experimental): Providing treatment as usual (detoxificaion) & psychotherapy
  Interventions: Behavioral: Detoxification & psychotherapeutic support

INTERVENTIONS:
Behavioral: Detoxification & psychotherapeutic support

SUMMARY:
The aim of the study is to evaluate effectiveness of inpatient detoxification and psycho-therapeutic support, measured in terms of readiness to change and abstinence maintenance. The study participants will be the patients admitted for alcohol use disorder (age: 18 years above) at a tertiary level hospital in Kathmandu. Baseline assessments on readiness to change will be done during admission, and compared prior to and after discharge. Percentage of participants maintaining abstinence in 3 months after discharge will be another outcome to be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as ADS according to ICD 10

Exclusion Criteria:

* Major Psychiatric or medical comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) Short Form | Change from baseline at discharge, an average of 2 weeks
  The questionnaire is 19 item self-report questionnaire assessing client readiness for change. There are three sub scales: Recognition, Ambivalence, and Taking Steps. Higher scores indicate greater recognition, ambivalence and taking steps. Scores range from 7 to 35, 4 to 20, and 8-40, respectively.
Percentage of participants staying abstinent | Three month follow up
  Percentage of participants not taking single drink or staying complete abstinent

IPD SHARING:
Plan to Share IPD: Undecided
If required, it will be discussed among the team and will be decided on need basis